CLINICAL TRIAL: NCT06564961
Title: The Effect of Clomiphene Citrate on Sperm Parameters in Infertile Men With Idiopathic Oligoasthenozoospermia
Brief Title: Clomiphene Citrate in Infertile Men With Idiopathic Oligoasthenozoospermia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shakeela Ishrat (Other)
Responsible Party: Sponsor-Investigator, Shakeela Ishrat, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Organization: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4068
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Male
Keywords: Male infertility; Oligoasthenozoospermia; Testosterone; Clomiphene citrate
MeSH Terms: conditions — Infertility, Male | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clomiphene (Experimental): Participants will receive Tab Clomiphene citrate 50 mg orally once daily or 12 weeks
  Interventions: Drug: Clomiphene Citrate
- Placebo (Placebo Comparator): Participants will receive Clomiphene citrate placebo tablet matching Clomiphene citrate orally once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clomiphene Citrate — 50 mg tab once daily
  Other Names: Tab OVULET (Renata Pharmaceuticals Limited)
  Arms: Clomiphene
Drug: Placebo — 1 tab once daily
  Other Names: Placebo provided by Renata Pharmaceuticals Limited
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug clomiphene citrate improves sperm parameters in infertile men with idiopathic oligoasthenozoospermia. It will also learn about the safety of clomiphene citrate. The main questions it aims to answer are:

* Does drug clomiphene citrate change sperm count and motility in infertile men with idiopathic oligoasthenozoospermia?
* What medical problems do participants have when taking drug clomiphene citrate? Researchers will compare drug clomiphene citrate to a placebo (a look-alike substance that contains no drug) to see if drug clomiphene citrate works to treat idiopathic oligoasthenozoospermia.

ELIGIBILITY:
Inclusion Criteria:

* Infertile men
* Idiopathic oligoasthenozoospermia (serum FSH and serum LH range was 2-7 IU/mL and serum testosterone level was >300 ng/dl)

Exclusion Criteria:

* Azoospermia
* Body mass index <18 kg/m2 and >30 kg/m2
* Any abnormality on genital examination and scrotal sonogram
* History of genital diseases & genital surgery
* Medical and endocrine disorders like uncontrolled diabetes mellitus, severe kidney disease and liver insufficiency
* Psycho-sexual abnormalities
* Antioxidant supplements in previous 3 months
* Smoking, drug, alcohol or substance abuse
* History of chemotherapy or radiotherapy
* Presence of any gross female factor abnormality

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 50 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sperm motility at 12 weeks | Baseline and 12 weeks
  Sperm motility was percentage of progressive & non-progressive motility
Change from baseline in sperm count at 12 weeks | Baseline and 12 weeks
  Sperm count was in million per milliliter of semen

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chehab M, Madala A, Trussell JC. On-label and off-label drugs used in the treatment of male infertility. Fertil Steril. 2015 Mar;103(3):595-604. doi: 10.1016/j.fertnstert.2014.12.122. Epub 2015 Feb 3. PMID 25660648
- [Background] Jung JH, Seo JT. Empirical medical therapy in idiopathic male infertility: Promise or panacea? Clin Exp Reprod Med. 2014 Sep;41(3):108-14. doi: 10.5653/cerm.2014.41.3.108. Epub 2014 Sep 30. PMID 25309854
- [Background] Cocuzza M, Agarwal A. Nonsurgical treatment of male infertility: specific and empiric therapy. Biologics. 2007 Sep;1(3):259-69. PMID 19707335
- [Background] Chua ME, Escusa KG, Luna S, Tapia LC, Dofitas B, Morales M. Revisiting oestrogen antagonists (clomiphene or tamoxifen) as medical empiric therapy for idiopathic male infertility: a meta-analysis. Andrology. 2013 Sep;1(5):749-57. doi: 10.1111/j.2047-2927.2013.00107.x. PMID 23970453
- [Background] Bridges N, Trofimenko V, Fields S, Carrell D, Aston K, Hotaling J. Male Factor Infertility and Clomiphene Citrate: A Meta-Analysis-The Effect of Clomiphene Citrate on Oligospermia. Urol Pract. 2015 Jul;2(4):199-205. doi: 10.1016/j.urpr.2014.10.007. Epub 2015 Apr 10. PMID 37559276
- [Background] Huijben M, Huijsmans RLN, Lock MTWT, de Kemp VF, de Kort LMO, van Breda JHMK. Clomiphene citrate for male infertility: A systematic review and meta-analysis. Andrology. 2023 Sep;11(6):987-996. doi: 10.1111/andr.13388. Epub 2023 Jan 29. PMID 36680549
- [Result] ElSheikh MG, Hosny MB, Elshenoufy A, Elghamrawi H, Fayad A, Abdelrahman S. Combination of vitamin E and clomiphene citrate in treating patients with idiopathic oligoasthenozoospermia: A prospective, randomized trial. Andrology. 2015 Sep;3(5):864-7. doi: 10.1111/andr.12086. Epub 2015 Jul 31. PMID 26235968